CLINICAL TRIAL: NCT03241927
Title: A Phase II Study Assessing the Effect of Pembrolizumab Induced Changes to the NK Cell Exhaustion Phenotype on the Efficacy of PD-1 Targeted Treatment in Patients With Unresectable Stage III or Stage IV Melanoma
Brief Title: Pembrolizumab Effects on NK Cell Exhaustion in Melanoma (Merck NK-IIT)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: difficult enrollment
Sponsor: Nina Bhardwaj (Other)
Responsible Party: Sponsor-Investigator, Nina Bhardwaj, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-2526
Record Dates: First submitted 2017-08-02; First posted 2017-08-08 (Actual); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Melanoma
Keywords: Pembrolizumab; NK Cell Exhaustion; PD-1; Unresectable; Stage III; Stage IV
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): 200 mg IV infusion every 3 weeks
  Interventions: Biological: Pembrolizumab
- Healthy Donors (No Intervention)

INTERVENTIONS:
Biological: Pembrolizumab — Day 1 of each 3 week cycle
  Arms: Pembrolizumab

SUMMARY:
Melanoma is an immune-modulated malignancy and immune checkpoint modulators which inhibit PD-1 function (pembrolizumab, nivolumab) have demonstrated clinical efficacy as treatment for patients with stage IV melanoma. Pembrolizumab across a range of doses in phase I investigation has demonstrated clinical efficacy with RR approximately 27%. By better understanding how NK cell function and exhaustion interplays with PD1 function and activity, potentially more efficacious combination therapies can be developed. The pharmacodynamic studies to be performed as part of this trial will provide such information.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Have Unresectable stage III or stage IV melanoma
* Be ≥ 18 years of age on day of signing informed consent.
* Have measurable disease based on RECIST 1.1 and be able to be followed over time by Immune related response criteria (irRC) for treatment decisions.
* Have a performance status of 0, 1, or 2 on the ECOG Performance Scale.
* Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.
* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.6.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of systemic immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Topical, inhaled, ocular, and intra-articular steroids are not exclusionary.
* Has a known history of active TB (Bacillus Tuberculosis).
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) treatment within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. - Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
* Note: If subject received major surgery, the subject must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided the subjects are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* If pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.
* Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bhardwaj, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 Participants consented, 1 with unstable CNS and not eligible, 2 withdrew consent. and 1 enrolled.
Groups:
- Healthy Donors: Healthy participants
Period: Overall Study
Arm/Group | Pembrolizumab | Healthy Donors
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — study terminated | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 1
Age, Customized [Count of Participants; unit: Participants]
  60-69 years | 1
  70-79 years | 0
  80-89 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent of LAMP-1 Positive Cells
Description: NK cell exhaustion will be assess by flow cytometry and expressed as % of LAMP-1 positive cells.
Time Frame: up to 3 years
Population: Data not collected
Arm/Group | Pembrolizumab | Healthy Donors
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Percent of Positive Cell for IFN Gamma
Description: IFN gamma will be assess by flow cytometry and then expressed as % of positive cell for IFN gamma.
Time Frame: up to 3 years
Population: Data not collected
Arm/Group | Pembrolizumab | Healthy Donors
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Percent of Proliferating Cells
Description: NK proliferation will be assess by flow cytometry and then expressed as percentage of proliferating cells.
Time Frame: up to 3 years
Population: Data not collected
Arm/Group | Pembrolizumab | Healthy Donors
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: MICA Plasma Level
Description: MICA plasma biomarker level associated with reversal of NK cell exhaustion will be assessed by ELISA.
Time Frame: up to 104 levels
Population: Data not collected
Arm/Group | Pembrolizumab | Healthy Donors
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: HMGB-1 Plasma Level
Description: HMGB-1 plasma biomarker level associated with reversal of NK cell exhaustion will be assessed by ELISA.
Time Frame: up to 104 weeks
Population: Data not collected
Arm/Group | Pembrolizumab | Healthy Donors
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: % of Positive NK Cells for CEACAM-1
Description: CEACAM-1 expression will be assessed by flow cytometry and express as % of positive NK cells for CEACAM-1
Time Frame: up to 104 weeks
Population: Data not collected
Arm/Group | Pembrolizumab | Healthy Donors
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Incidence of Overall Survival
Description: One year survival following pembrolizumab treatment in patients with Unresectable stage III or IV melanoma using Immune-Related Response Criteria.
Time Frame: 1 year
Population: Data not collected
Arm/Group | Pembrolizumab | Healthy Donors
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Progression Free Survival (PFS) Rate
Description: Progression free survival in pembrolizumab treated patients with unresectable stage III or IV melanoma using Immune-Related Response Criteria.
Time Frame: 6 months
Population: only one subject in study
Measure: Number; unit: weeks
Arm/Group | Pembrolizumab | Healthy Donors
Number analyzed (Participants) | 1 | 0
weeks | 18 |

ADVERSE EVENTS:
Time Frame: 18 weeks
Description: there was only one person in this study. No participants in Healthy Control arm.
Groups:
- Healthy Control: Healthy Participants
Arm/Group | Pembrolizumab | Healthy Control
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=1) | Healthy Control (N=0)
Bilateral Leg Edema (General disorders) | 1 (1) | 0
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Anemia (Blood and lymphatic system disorders) | 1 (3) | 0
Creatinine Increased (Investigations) | 1 (1) | 0
Hair thinning (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2) | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/27/NCT03241927/Prot_SAP_000.pdf